CLINICAL TRIAL: NCT07359196
Title: Assessment of Carbohydrate Content Estimation Among Sohag University Students With Type 1 Diabetes Mellitus and Their Glycemic Control
Brief Title: Assessment of Carbohydrate Counting Accuracy and Glycemic Control Among Sohag University Students With Type 1 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elzahraa Abdellatif Mohamed, Assistant Lecturer of Family Medicine, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-12-10MD
Record Dates: First submitted 2026-01-01; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: HA1c; Glycemic control; Nutrition education; PedCarbQuiz; Carbohydrate counting
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational intervention ( knowledge) (Experimental): Participants receiving carbohydrate counting education.
  Interventions: Behavioral: Carbohydrate Counting Education

INTERVENTIONS:
Behavioral: Carbohydrate Counting Education — educational session on carbohydrate counting and insulin dose adjustment.

SUMMARY:
This study assesses carbohydrate counting knowledge and its impact on glycemic control among Sohag University students with type 1 diabetes mellitus. A structured educational intervention will be delivered, followed by reassessment after three months.

DETAILED DESCRIPTION:
This interventional study targets undergraduate students diagnosed with type 1 diabetes mellitus at Sohag University. Baseline data will include demographic characteristics, diabetes-related history, carbohydrate counting knowledge assessed using the PedCarbQuiz, and glycemic control parameters including HbA1c.

Participants will receive a structured educational session focusing on carbohydrate counting principles and insulin dose adjustment. Educational booklets will be provided. After three months, carbohydrate counting knowledge and glycemic control will be reassessed to evaluate the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of T1DM for at least 1 year.
2. Age ≥18 years.
3. Currently enrolled at Sohag University.
4. Willing to participate and provide informed consent.

Exclusion Criteria:

1. University students who refuse to participate in the study
2. Students with other types of diabetes (T2DM, MODY, etc.)
3. Presence of other chronic illnesses that affect diet or glycemic control (e.g., celiac disease, chronic kidney disease).
4. Students with communication barriers e.g cognitive impairment or psychiatric illness interfering with questionnaire completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c | 3 months

SECONDARY OUTCOMES:
Change in Carbohydrate counting knowledge | base line and 3 months
  Using PedCarbQuiz

IPD SHARING:
Plan to Share IPD: Undecided